CLINICAL TRIAL: NCT02359084
Title: Early Identification and Service Linkage for Urban Children With Autism
Brief Title: Project EARLY: Engagement, Assessment, Referral, & Linkage for Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Yale University (Other); Children's Hospital of Philadelphia (Other); National Institute of Mental Health (NIMH) (NIH); Developmental Behavioral Pediatrics Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: H-33008; 1R01MH104355 (NIH)
Record Dates: First submitted 2015-02-01; First posted 2015-02-09 (Estimated); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Autism; Developmental Delay Disorders
Keywords: Autism Spectrum Disorder (ASD); Family navigation
MeSH Terms: conditions — Autistic Disorder; Developmental Disabilities; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Navigation (Experimental): Families will work one-on-one with the navigator who provides off-site support - e.g. home visits or accompanying families to appointments. The goal of FN during the diagnostic evaluation period is to ensure timely completion of the evaluation. The focus of these interactions is to understand the structure and purpose of the evaluation, gather and complete required materials, and address logistic barriers related to the diagnostic visit. The navigator will continue to work with the family after the diagnostic evaluation to access recommended services and support the family's engagement in treatment.
  Interventions: Behavioral: Family Navigation
- Conventional Care Management (Active Comparator): Families will be assigned to a care manager for the diagnostic evaluation and for 100 days thereafter. Consistent with a high quality medical home, the care manager will be responsible to ensure that the referral for the diagnostic evaluation has been made. She is also available for family-initiated support. The care manager will be responsible for ensuring that referrals are made and continue to provide family-initiated, clinic-based support to families for up to 100 days after the completion of diagnostic evaluation.
  Interventions: Behavioral: Conventional Care Management

INTERVENTIONS:
Behavioral: Family Navigation
  Arms: Family Navigation
Behavioral: Conventional Care Management
  Arms: Conventional Care Management

SUMMARY:
Emerging evidence demonstrates that Autism Spectrum Disorder (ASD) can be reliably diagnosed by age two, and that early identification and intervention can improve outcomes. Low-income and minority children with ASD, however, are diagnosed later and experience greater delays in service provision than their white and more financially advantaged peers. Feasible, culturally appropriate interventions with broad scale-up potential are necessary to reduce this disparity. This project builds upon pilot studies of an adapted version of Patient Navigation, as means to reduce disparities in ASD diagnosis and service provision. Patient Navigation is a lay-delivered case management approach that focuses on overcoming logistical hurdles to care during a defined episode.

This project has 2 components, both of which take place in urban, integrated care networks that provide healthcare to low-income children. This registration is for the clinical trial component of the study. The project is a multisite, randomized comparative effectiveness trial of a systemic, lay-delivered adaptation of Patient Navigation, referred to as Family Navigation (FN), which begins with a failed autism screen and ends 100 days after an ASD diagnosis is made. The basic structure of both intervention arms is a collaborative care system. The conventional care management arm (CCM) is consistent with the type of care provided within a traditional - but high quality - medical home. The FN arm provides more intensive, individually tailored, care coordination and theory-based family support.

DETAILED DESCRIPTION:
We will conduct a randomized, comparative effectiveness trial to test a systemic, lay-delivered FN protocol against conventional care management services. The study will take place in three integrated primary care networks and their affiliated Developmental and Behavioral Pediatrics (DBP) clinics at Boston Medical Center, Children's Hospital of Philadelphia, and Yale University Medical School. We will enroll children with confirmed risk for ASD in the randomized trial and will employ 1:1 randomization by child. The FN protocol will include individualized navigation to support completion of the diagnostic evaluation, referral to appropriate services, and linkage to and engagement in services. We will determine FN's effect on identifying children at risk for ASD, timing of diagnosis, and receipt of evidence-based ASD services.

The study seeks to accomplish the following aims:

1. Implement a decision rule for referral for formal ASD evaluation;
2. Ensure timely diagnosis and deployment of services.

If successful, our study will provide real world primary care practices with a replicable model of care that increases early identification and access to timely diagnostic and early intervention services for a vulnerable population of urban families.

Children will be followed for 12 months. Data regarding screening outcomes, diagnosis and service utilization will be abstracted from children's medical records. Measures of parental stress, self-management skills, caregiver burden, and satisfaction with services will be administered over 4 collection time points, linked to key intervention outcomes. We will assess the superiority of FN as compared to CCM as a means to: implement a decision rule for referral to ASD evaluation; shorten the time to diagnosis among children suspected to have ASD; shorten the time to deployment of ASD services among those diagnosed; and improve engagement with ASD services.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 15 - 27 months at a participating clinic who fail the M-CHAT screen and/or primary care provider has concerns about autism

Exclusion Criteria:

* Previous diagnosis of Autism Spectrum Disorder

Ages: 15 Months to 27 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 340 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic interval (Number of days defined as beginning the day of the positive confirmatory screen and ending the day when the family receives a determination (yes/no) of ASD diagnosis) | On average 90 -120 days, specific date is linked to the completion of the developmental assessment
  Number of days defined as beginning the day of the positive confirmatory screen and ending the day when the family receives a determination (yes/no) of ASD diagnosis
Time to receipt of ASD services/recommended services | 1 year
  Number of days from date of diagnosis to receipt of recommended services

SECONDARY OUTCOMES:
Determination of ASD diagnosis (based on DSM V criteria made by a Board Certified DBP Pediatrician. Assessments are based on site protocols; all use standardized, validated measures appropriate for very young children.) | 1 year
  Determination of ASD diagnosis will be based on DSM V criteria made by a Board Certified DBP Pediatrician. Assessments are based on site protocols; all use standardized, validated measures appropriate for very young children.
Satisfaction with Family Navigator (Patient Satisfaction with Interpersonal Relationship with Navigator (PSN-I)) | 100 days after developmental assessment completion
  Patient Satisfaction with Interpersonal Relationship with Navigator (PSN-I) is a newly validated 9 item scale to assess satisfaction with the interpersonal relationship with the navigator.

OTHER OUTCOMES:
Perceived Stress Scale - Self Report | 1-4 weeks after developmental assessment completion, 100 days after developmental assessment completion, 1 year after failed confirmatory screen
  The Perceived STress Scale is a measure of the degree to which situations in one's life are appraised as stressful. The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way.; lower scores are more favorable.
Parenting Stress Index - Short Form | 1-4 weeks after developmental assessment completion, 100 days after developmental assessment completion, 1 year after failed confirmatory screen
  This measure is a brief version of the Parenting Stress Index, a widely used and well-researched measure of parenting stress. The PSI-SF has 36 items from the original 120-item PSI. Items are identical to those in the original version. It was developed in response to clinicians' and researchers' need for a shorter measure of parenting stress and was based on Castaldi's factor analysis of the original PSI, which suggested the presence of three factors. It yields scores on the following subscales: 1) Parental Distress, 2) Parent-Child Dysfunctional Interaction, and 3) Difficult Child. Similar to the full PSI, it also has a validity scale.
Brief COPE | 1-4 weeks after developmental assessment completion, 100 days after developmental assessment completion, 1 year after failed confirmatory screen
Pearlin Mastery Scale | 1-4 weeks after developmental assessment completion, 100 days after developmental assessment completion, 1 year after failed confirmatory screen
  The Pearlin Mastery Scale is designed to measure self-concept and references the extent to which individuals perceive themselves in control of forces that significantly impact their lives. Total score can range from 7 to 28 points; higher scores are more favorable.
VR12 Health Survey | 1-4 weeks after developmental assessment completion, 100 days after developmental assessment completion, 1 year after failed confirmatory screen
  VR-12 includes 12 original question items from the VR-36. The questions in this survey correspond to seven different health domains: general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy/fatigue levels, social functioning and mental health.
MOS-Social Support Survey | 1-4 weeks after developmental assessment completion, 100 days after developmental assessment completion, 1 year after failed confirmatory screen
  This is a brief, multidimensional, self-administered, social support survey that was developed for patients in the Medical Outcomes Study (MOS), a two-year study of patients with chronic conditions. This survey was designed to be comprehensive in terms of recent thinking about the various dimensions of social support.
Family Impact Questionnaire | 1-4 weeks after developmental assessment completion, 100 days after developmental assessment completion, 1 year after failed confirmatory screen
Autism Parenting Stress Index (APSI) | 1-4 weeks after developmental assessment completion, 100 days after developmental assessment completion, 1 year after failed confirmatory screen
  Screening and triage measure for evaluating the parenting system and identifying issues that may lead to problems in the child's or parent's behavior. Focuses on three major domains of stress: child characteristics, parent characteristics and situational/demographic life stress.
Adaptive Behavior Assessment System | 1 year after failed confirmatory screen
  Communication, Social, and Self-Direction subscales
Brief Illness Perception Questionnaire | 1 year after failed confirmatory screen
Hospital Care Questionnaire | 100 days after developmental assessment completion, 1 year after failed confirmatory screen
Engagement in treatment | 1 year
  Number of hours of ASD/general developmental services
Mullen Scales of Early Learning (MSEL) | 1 year after failed confirmatory screen
  Visual Reception, Fine Motor, Receptive Language, and Expressive Language scales
Vineland Adaptive Behavior Scales-3 | 1 year after failed confirmatory screen
  Parent/caregiver rating form; all domains except motor and maladaptive
Autism Diagnostic Observation Schedule-2 | at time of evaluation and 1 year after failed confirmatory screen

CONTACTS AND LOCATIONS:
Overall Officials: Emily Feinberg, ScD, Principal Investigator — Boston University
Locations (10):
- United States (10):
  - Yale University School of Medicine, New Haven, Connecticut
  - Boston Medical Center, Boston, Massachusetts
  - Boston University School of Public Health, Boston, Massachusetts
  - South End Community Health Center, Boston, Massachusetts
  - Dorchester House Multi-Service Center, Boston, Massachusetts
  - Codman Square Health Center, Boston, Massachusetts
  - East Boston Neighborhood Health Center, Boston, Massachusetts
  - MGH Chelsea, Chelsea, Massachusetts
  - Lowell Community Health Center, Lowell, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the National Database for Autism Research biannually.

REFERENCES:
- [Derived] Levinson J, Hickey E, Fuchu P, Chu A, Barnett M, Stadnick NA, Feinberg E, Broder-Fingert S. Recommendations for post-implementation adaptations to optimize family navigation in pediatric primary care: a qualitative study with parents and navigators. BMC Prim Care. 2023 Jun 16;24(1):123. doi: 10.1186/s12875-023-02072-y. PMID 37328810
- [Derived] Eilenberg JS, Kizildag D, Blakey AO, Cardona ND, Oberoi A, Broder-Fingert S, Feinberg E, Long KA. Implications of Universal Autism Screening: Perspectives From Culturally Diverse Families With False-Positive Screens. Acad Pediatr. 2022 Mar;22(2):279-288. doi: 10.1016/j.acap.2021.12.025. Epub 2021 Dec 25. PMID 34963655
- [Derived] Feinberg E, Augustyn M, Broder-Fingert S, Bennett A, Weitzman C, Kuhn J, Hickey E, Chu A, Levinson J, Sandler Eilenberg J, Silverstein M, Cabral HJ, Patts G, Diaz-Linhart Y, Fernandez-Pastrana I, Rosenberg J, Miller JS, Guevara JP, Fenick AM, Blum NJ. Effect of Family Navigation on Diagnostic Ascertainment Among Children at Risk for Autism: A Randomized Clinical Trial From DBPNet. JAMA Pediatr. 2021 Mar 1;175(3):243-250. doi: 10.1001/jamapediatrics.2020.5218. PMID 33427861
- [Derived] Broder-Fingert S, Walls M, Augustyn M, Beidas R, Mandell D, Wiltsey-Stirman S, Silverstein M, Feinberg E. A hybrid type I randomized effectiveness-implementation trial of patient navigation to improve access to services for children with autism spectrum disorder. BMC Psychiatry. 2018 Mar 27;18(1):79. doi: 10.1186/s12888-018-1661-7. PMID 29587698